CLINICAL TRIAL: NCT05030051
Title: A Proof of Concept Study to Evaluate the Efficacy and Tolerability of Skinpen on Male and Female Subjects' Dorsal Hands as a Treatment of Hand Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crown Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-HAS-21-03
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SkinPen Precision System (Experimental): This proof of concept study is being conducted over the course of 60 days followed by a 3-month post-treatment visit to assess the efficacy and tolerability of the Sponsor's SkinPen device when used to treat men and women with signs of aging on the dorsum of the hands. Overall assessment of clinical outcome and safety will be based on the evaluation of pre- and post-treatment photos comparing baseline to final visit. The subject's assessment of satisfaction will also be evaluated at Visit 3 and Visit 4. Finally, both the clinician's and subject's assessment will be characterized using a clinician assessment scale at the 3 month post-treatment visit.
  Interventions: Device: SkinPen Precision System

INTERVENTIONS:
Device: SkinPen Precision System — Microneedling is a relatively new, minimally invasive technique originally developed for skin rejuvenation. Controlled micro-injury to the dermis via the application of several small needles connected to a motorized device stimulates the wound healing process, resulting in the formation of new tissue and blood vessels. The SkinPen by Crown Laboratories is an FDA-cleared microneedling device proven to improve the appearance of acne scars This study evaluates the clinical performance of the SkinPen device for the treatment of signs of aging on the back of the hand. We hypothesize that the SkinPen device will produce a significant improvement in dorsal hand appearance at 3 month post treatment visit, when compared with baseline scores. The assessments will be based on the Clinician's Global Aesthetic Improvement Scale, and the Subject's Global Aesthetic Improvement Scale at the 3 month post treatment visit.

SUMMARY:
This proof of concept study is being conducted over the course of 60 days followed by a 3-month post-treatment visit to assess the efficacy and tolerability of the Sponsor's SkinPen device when used to treat men and women with signs of aging on the dorsum of the hands. Overall assessment of clinical outcome and safety will be based on the evaluation of pre-and post-treatment photos comparing baseline to final visit. The subject's assessment of satisfaction will also be evaluated at Visit 3 and Visit 4. Finally, both the clinician's and subject's assessments will be characterized using a clinician assessment scale at the 3-month post-treatment visit.

DETAILED DESCRIPTION:
A total of 18 subjects will be enrolled in this study. These patients will be treated three times over the dorsum of the hand from the wrist to the knuckles each month for three months, followed by one follow-up visit at 3-months post-treatment.

Blueberry and Crown Laboratories will be responsible for recruitment efforts. Subjects will be numbered sequentially in the order in which they qualify for entry into the study.

3.2 Primary Endpoints • Clinician's global aesthetic improvement assessment (CGAIS) at 3-months post-treatment.

3.3 Secondary Endpoints

* Subject's global aesthetic improvement assessment (SGAIS) at 3-months post-treatment.
* Monitoring of adverse events throughout the course of the study. Safety Subject diaries will be monitored for resolution of anticipated treatment responses.

3.4 Exploratory Endpoints

• Bioinstrumentation: TEWL, hydration, elasticity, skin thickness measurements at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 50 to 75 years of age in general good health.
* Individuals deemed by the Investigator, visually, to have signs of hand aging (presence of skin laxity, age spots, trophic changes) on the dorsum of the hand. Also, Subjects would have to be willing to undergo correction of these signs of aging.
* Individuals willing to withhold aesthetic therapies to the areas of the hand being treated or judged to potentially impact results by the Investigator (e.g. soft tissue fillers and/or any resurfacing procedures, botulinum toxin, injectable fillers, microdermabrasion, IPL (intense pulsed light), peels, laser treatments, and tightening treatments, etc.) for the duration of the study. Waxing and threading is allowed but not laser hair removal.
* Individuals that are willing to provide written informed consent.
* Individuals willing to sign a photography release.
* Willingness to cooperate and participate by following study requirements for the duration of the study and to report any changes in health status or medications, adverse event symptoms, or reactions immediately.
* Women of childbearing potential agree to take a urine pregnancy test at the Baseline visit and 3-months post-treatment or when deemed by Investigator and/or Sponsor. This may be changed to a monthly pregnancy test at the Sponsor's discretion. Women who are of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the baseline visit. Women must be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

  * Postmenopausal for at least 12 months prior to study.
  * Without a uterus and/or both ovaries.
  * Bilateral tubal ligation at least 6 months prior to study enrollment
* Exclusion Criteria:
* Individuals diagnosed with known allergies to general skin care products.
* Individuals who have presence of an active systemic or local skin disease that may affect wound healing.
* Individuals with sensitivity to topical lidocaine.
* Individuals who have physical or psychological conditions unacceptable to the Investigator.
* Individuals who have a recent history of significant trauma to the areas to be treated (< 6 months).
* Individuals who have significant scarring in the area(s) to be treated.
* Individuals who have a recent or current history of inflammatory skin disease, infection or unhealed wound.
* Individuals who have a history of systemic granulomatous diseases, active or inactive, (e.g. Sarcoid, Wegeners, TB, etc.) or connective tissue diseases (e.g. lupus, dermatomyositis, etc.).
* Individuals who currently have or have a history of hypertrophic scars, or keloid scars.
* Individuals who currently have cancerous or pre-cancerous lesions in the areas to be treated and/or with a history of skin cancer.
* Individuals who have the inability to understand instructions or to give informed consent.
* Individuals who have had microdermabrasion or glycolic acid treatment to the treatment area(s) within one month prior to study participation or who will have this treatment during the study.
* Individuals who have a history of chronic drug or alcohol abuse.
* Individuals undergoing concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Individuals who, in the Investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Individuals who are current smokers.
* Individuals who have a history of the following cosmetic treatments in the area(s) to be treated:

  * Skin tightening procedure within the past year;
  * Injectable filler of any type within the past:
* 12 months for Hyaluronic acid fillers (e.g. Restylane)
* 12 months for Ca Hydroxyapatite fillers (e.g. Radiesse)
* 24 months for Poly-L-Lactic acid fillers (e.g. Sculptra)
* Ever for permanent fillers (e.g. Silicone, ArteFill)

  * Ablative resurfacing laser treatment;
  * Non-ablative, rejuvenative laser or light treatment within the past six months;
  * Surgical dermabrasion;
  * Had a chemical peel or dermabrasion, of the dorsum of the hand within four weeks
* Individuals with a history of using the following prescription medications:

  * Accutane or other systemic retinoids within the past six months;
  * Topical Retinoids within the past two weeks;
  * Prescription strength skin lightening devices (e.g. hydroquinone, tretinoin, AHA, BHA and polyhydroxy acids, 4-hydroxyanisole alone or in combination with tretinoin, etc.) within four months;
  * Any anti-wrinkle, skin lightening devices, or any other device or topical or systemic medication known to affect skin aging or dyshcromia (devices containing alpha/beta/poly-hydroxy acids, vitamin C, soy, Q-10, hydroquinone; systemic or licorice extract (topically), Tego® Cosmo C250, gigawhite, lemon juice extract (topically), emblica extract, etc.) within two weeks;
  * Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix, chronic NSAID use); and/or
  * Psychiatric drugs that in the Investigator's opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.
* Individuals who are nursing, pregnant, or planning to become pregnant during the study according to subject self-report.
* Individuals having a health condition and/or pre-existing or dormant dermatologic disease on the body (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation) that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
* Individuals with a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) and/or radiation as determined by study documentation.
* Individuals with an uncontrolled disease such as asthma, diabetes, hyperthyroidism, medically significant hypertension or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
* Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures during the course of the study.
* Individuals who have observable suntan, nevi, excessive hair, etc. or other dermal conditions on the back of the hand that might influence the test results in the opinion of the Investigator or designee.
* Individuals who have any condition, which in the opinion of the Investigator makes the patient unable to complete the study per protocol (e.g. patients not likely to avoid other cosmetic treatments to the treatment area; patients not likely to stay in the study for its duration because of other commitments, concomitant conditions, or past history; patients anticipated to be unreliable, or patients who have a concomitant condition that may develop symptoms that might confuse or confound study treatments or assessments).
* Individuals who started hormone replacement therapies (HRT) or hormones for birth control less than three months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Clinician's global aesthetic improvement assessment (CGAIS) | 3-Month Post Treatment
  This scale should be completed:
  • Based on a live assessment of the subject while referring to the subject's pre-treatment photographs of the dorsal hand and final visit
  Rating Description
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re-treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.

SECONDARY OUTCOMES:
Subject's global aesthetic improvement assessment (SGAIS) | 3-Month Post Treatment
  At final visit, Subjects will be presented with Baseline and Visit 4 Photographs to complete this assessment.
  Rating Description
  1. Very Much Improved: Optimal cosmetic result.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal.
  3. Improved: Obvious improvement in appearance from initial condition.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Crown Laboratories, Dallas, Texas, United States